CLINICAL TRIAL: NCT01918683
Title: A Pilot Trial of Transarterial Chemoembolization With or Without Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma Patients Awaiting Liver Transplantation
Brief Title: TACE With or Without SBRT as Bridging Therapy for Pre-transplant HCC Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Loyola University (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 16213
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: two arms
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A -Tace alone (Other): A - TACE alone (control group, current practice and treatment)
  Interventions: Radiation: TACE transarterial chemoembolization
- B - Tace combined with SBRT (Experimental): B- TACE combined with SBRT (experimental group).
  Interventions: Radiation: TACE transarterial chemoembolization; Radiation: stereotatic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: TACE transarterial chemoembolization
Radiation: stereotatic body radiotherapy (SBRT)
  Arms: B - Tace combined with SBRT

SUMMARY:
This trial is designed to be the initial prospective pilot investigation of the effectiveness of combined SBRT and TACE as bridging therapy for HCC patients awaiting liver transplanation. No prospective clinical trials regarding the combination of TACE and SBRT in pre-transplant population have been performed. We propose the trial be conducted as a pilot clinical trial with the goal of enrolling 40 patients into each arm

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the combination of stereotatic body radiotherapy (SBRT) tand transarterial chemoembolization (TACE) is an effective "bridging therapy" for patients hepatocellular carcinoma (HCC) of the liver awaiting transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of giving informed consent
* Patient diagnosed with hepatocellular carcinoma and listed or recommended to be listed for orthotopic liver transplantation at the participating institution
* Age > 18 years old
* Meets clinical criteria for eligibility for TACE to the target lesion per Interventional Radiology
* Childs' Class A or B7
* Eastern Clinical Oncology Group performance status 0 or 1

Exclusion Criteria:

* Prior radiotherapy to the upper abdomen or radioembolization of the liver
* Prior TACE to the target lesion, RFA, or liver transplant
* Active GI bleed within 2 weeks of study enrollment
* Active GI ulcer disease within 4 weeks of study enrollment
* Ascites refractory to medical therapy
* Contraindication to receiving radiotherapy or TACE
* Complete obstruction of portal venous flow to the segment of liver that includes the target lesion
* Contraindication to both contrast enhanced MRI and contrast enhanced CT (i.e. unable to undergo follow-up imaging or SBRT treatment planning)
* Women who are pregnant
* Participation in another concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-07; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 10 days
  endpoint is OLT

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Ben-Josef, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Tarita Thomas, MD, PhD, Principal Investigator — Loyola University
Locations (3):
- United States (3):
  - Loyola University Medical Center, Maywood, Illinois
  - Oregon Health & Science University, Portland, Oregon
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania